CLINICAL TRIAL: NCT05200221
Title: A Single Center Real-world Study of Donafenib in the Treatment of Hepatocellular Carcinoma (HCC) in Routine Clinical Practice
Brief Title: A Single Center Real-world Study of Donafenib in the Treatment of Hepatocellular Carcinoma in Routine Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-569R
Record Dates: First submitted 2022-01-17; First posted 2022-01-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Donafenib; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Donafenib: Patients with uHCC taking donafenib in clinical treatment

SUMMARY:
This trial is a single center observational real-world study. It is planned to include 300 patients with unresectable hepatocellular carcinoma (uHCC) treated with Donafenib. The purpose of the study was to observe the effectiveness and safety of Donafenib in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Histologically confirmed HCC or meet the clinical diagnostic criteria of HCC;
3. Unresectable HCC;
4. The doctor decided to use donafenib before the patient was enrolled in the study；
5. Informed consent and willing to complete the study according to the protocol.

Exclusion Criteria:

1. Those who are participating in clinical trials of other antitumor drugs;
2. Allergic to any component of Donafenib tablets;
3. Patients with active bleeding, active peptic ulcer, drug uncontrollable hypertension or severe liver dysfunction;
4. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include 300 patients with unresectable hepatocellular carcinoma treated with Donafenib.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events. | an average of 1.5 year.
  Incidence of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Objective response rate (ORR) | an average of 1 year.
  According to RECIST v1.1 and mRECIST to evaluate the proportion of patients with complete response(CR) and partial response(PR) in the total number of patients.
Duration of remission (DoR) | an average of 1 year.
  Time from the date of first confirmed CR or PR to the occurrence of disease progression.
Disease control rate (DCR) | an average of 1 year
  According to RECIST v1.1 and mRECIST to evaluate the proportion of patients with CR, PR and stable disease(SD) in the total number of patients.
Progression-free survival(PFS) | an average of 1 year
  PFS refers to the time from the date of enrollment to tumor progression or death from any cause.
overall survival(OS) | an average of 1 year
  The time from the date of enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, M.D., Ph.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China.
Locations (1):
- Zhongshan Hospital, Fudan University,, Shanghai, Shanghai Municipality, China